CLINICAL TRIAL: NCT02079181
Title: 18F-FMAU for Imaging in Cancer Patients
Brief Title: 18F-FMAU PET/CT in Imaging Patients With Advanced Cancers
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Drug not available
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 0S-12-3; NCI-2014-00314 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 0S-12-3 (Other: USC Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2014-03-03; First posted 2014-03-05 (Estimated); Last update posted 2024-05-24 (Actual); Status verified 2023-08

CONDITIONS: Malignant Neoplasm
MeSH Terms: conditions — Neoplasms | interventions — clevudine; Magnetic Resonance Spectroscopy; 2-phenyl-6-(2'-(4'-(ethoxycarbonyl)thiazolyl))thiazolo(3,2-b)(1,2,4)triazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Diagnostic (fluorine F 18 d-FMAU PET/CT scan) (Experimental): Patients receive fluorine F 18 d-FMAU IV followed by PET/CT prior to start of cancer treatment. Patients may undergo 2 additional scans at one week prior to second course of chemotherapy and after completion of cancer treatment depending on cancer type.
  Interventions: Radiation: fluorine F 18 d-FMAU; Procedure: positron emission tomography; Procedure: computed tomography

INTERVENTIONS:
Radiation: fluorine F 18 d-FMAU — Given IV
Procedure: positron emission tomography — Undergo fluorine F 18 d-FMAU PET/CT scan
  Other Names: FDG-PET; PET; PET scan; tomography, emission computed
Procedure: computed tomography — Undergo fluorine F 18 d-FMAU PET/CT scan
  Other Names: tomography, computed

SUMMARY:
This clinical trial studies the safety and drug distribution of the radioactive drug, 2'-deoxy-2'-[18F]fluoro-5-methyl-1-beta-D-arabinofuranosyluracil (fluorine F 18 d-FMAU [18F-FMAU]), for imaging with positron emission tomography/computed tomography (PET/CT) in patients with advanced cancers. A PET scan is a procedure in which a small amount of radioactive glucose (sugar) is injected into a vein, and a scanner is used to make detailed, computerized pictures of areas inside the body where the glucose is taken up. Because cancer cells often take up more glucose than normal cells, the pictures can be used to find cancer cells in the body. PET/CT using the drug fluorine F 18 d-FMAU, may help find cancer and find out how far the disease has spread.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the radiation dosimetry of 18F-FMAU in humans, confirm absence of adverse events in humans from intravenous (i.v.) injection of 18F-FMAU for PET imaging, and characterize the incidence of circulating metabolites of 18F-FMAU in humans.

II. To simply find out whether there is any visual uptake change of 18F-FMAU in tumors post-therapy.

OUTLINE:

Patients receive fluorine F 18 d-FMAU IV followed by PET/CT prior to start of cancer treatment. Patients may undergo 2 additional scans at one week prior to second course of chemotherapy and after completion of cancer treatment depending on cancer type.

ELIGIBILITY:
Inclusion Criteria:

* Have been diagnosed with a malignancy/tumor/cancer, including but not limited to: brain tumor, breast cancer, lung cancer, esophageal cancer, lymphoma, or sarcoma
* Have one or more tumors visualized by conventional PET-CT, CT or magnetic resonance imaging (MRI) prior to the PET FMAU study; PET-CT should be within one week prior to 18F-FMAU

Exclusion Criteria:

* Have undergone chemotherapy or radiation therapy within the previous one month
* Women of childbearing potential, unless they have had a negative urine beta human chorionic gonadotropin (betaHCG) within the previous 24 hours of the procedure
* Patients who have had surgery at the site of the suspected lesion within 1 month

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2014-01-31 (Actual); Primary Completion 2023-08-22 (Actual); Study Completion 2023-08-22 (Actual)

PRIMARY OUTCOMES:
Radiation dosimetry of fluorine F 18 d-FMAU | Up to 24 hours after fluorine F 18 d-FMAU PET/CT scan
Adverse events after injection of fluorine F 18 d-FMAU to the patients | Up to 24 hours after fluorine F 18 d-FMAU PET/CT scan
Fluorine F 18 d-FMAU uptake change in tumors post-therapy | Baseline up to 24 hours after fluorine F 18 d-FMAU PET/CT scan

CONTACTS AND LOCATIONS:
Overall Officials: Peter Conti, MD, Principal Investigator — University of Southern California
Locations (1):
- USC Norris Comprehensive Cancer Center, Los Angeles, California, United States